CLINICAL TRIAL: NCT05713292
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Pirfenidone in Adult Hospitalized Patients With COVID-19.
Brief Title: Pirfenidone in Adult Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-China Pirfenidone
Record Dates: First submitted 2023-01-01; First posted 2023-02-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone (Experimental): Pirfenidone 200mg tid for first week; subsequently, 400mg tid for 2 months
  Interventions: Drug: Pirfenidone Oral Product
- Placebo (Placebo Comparator): Pirfenidone placebo 200mg tid for first week; subsequently, 400mg tid for 2 months
  Interventions: Drug: Pirfenidone placebo

INTERVENTIONS:
Drug: Pirfenidone Oral Product — Pirfenidone 200mg tid for first week; subsequently, 400mg tid for 2 months
  Arms: Pirfenidone
Drug: Pirfenidone placebo — Pirfenidone placebo
  Arms: Placebo

SUMMARY:
This center intends to conduct a multicenter, randomized, placebo-controlled study to evaluate the effectiveness and safety of Nintedanib ethanesulfonate soft capsule in the treatment of pulmonary fibrosis in patients with moderate to severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Age ≥ 18 Willing and able to provide written informed consent
* SARS-CoV-2 infection confirmed by PCR test/antigen dectection or positive serologies
* Time of illness onset ≥8 days
* Have findings consistent with interstitial lung disease found on CT scan
* Willing not use other investigational agents of anti-fibrosis

Exclusion Criteria:

* Pre-existing severe liver disease
* Pre-existing severe chronic kidney disease
* Pre-existing interstitial lung disease
* Pre-existing severe COPD or other structural lung disease
* Receiving invasive mechanical ventilation
* Currently Pregnant or Breast Feeding
* Poor baseline health conditoin
* Disability to complete lung function test
* Receiving pirfenidone wthin half-year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of pirfenidone on fibrotic signs induced by COVID19 infection | 1 month
  1. Change of total lung lesion volume on Chest CT from enrollment to 1 month follow up
  2. DLCO% pred at 1 month follow up

SECONDARY OUTCOMES:
distance walked in 6 Minutes (6MWD) | at the 1 month and 3 months follow-up vist
  the difference between intervention group and placebo group
the EuroQol five-dimension five-level (EQ-5D-5L) | at the 1 month and 3 months follow-up vist
  the difference between intervention group and placebo group
Medical Research Council (mMRC) dyspnoea scale | at the 1 month and 3 months follow-up vist
  the difference of mMRC score between intervention group and placebo group
difference of forced vital capacity (FVC) between two groups | at the 1 month and 3 months follow-up vist
  the difference of actual and predicted value between intervention group and placebo group
difference of total lung capacity (TLC) between two groups | at the 1 month and 3 months follow-up vist
  the difference of actual and predicted value between intervention group and placebo group
difference of DLCO between two groups | at the 3 months follow-up vist
  the difference of actual and predicted value between intervention group and placebo group
incidence of adverse event | within 2 months after enrollment
  the difference of adverse event frequency between intervention group and placebo group

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China